CLINICAL TRIAL: NCT06137937
Title: Intradialytic Aerobic Exercise in CKD Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Irma Ruslina Defi, Principal Investigator, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IKFR.10.23
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; intradialytic aerobic exercise; physical performance
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Thirty-four participants receiving hemodialysis were randomized to the intervention and control groups.
Masking Description: The sample in this study was determined randomly using a computer; subjects in the treatment group underwent routine hemodialysis by committing to an intradialysis aerobic exercise program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): subjects in the treatment group underwent routine hemodialysis by committing to an intradialysis aerobic exercise program
  Interventions: Behavioral: Aerobic Exercise
- Control Group (No Intervention): subjects in the control group underwent routine hemodialysis without a physical exercise program

INTERVENTIONS:
Behavioral: Aerobic Exercise — Intradialytic aerobic exercise for eight weeks
  Arms: Interventional Group

SUMMARY:
Intradialytic aerobic exercise is not effective in increasing hemodialysis adequacy but is effective in improving physical performance in twice-weekly hemodialysis patients.

DETAILED DESCRIPTION:
Uremic myopathy occurs in 60-75% of Chronic Kidney Disease (CKD) patients undergoing hemodialysis, which causes a decrease in muscle strength and physical performance. Increasing dialysis adequacy is beneficial in reducing the impact of uremia on muscles. Intradialytic aerobic exercise in thrice-weekly hemodialysis patients has improved dialysis adequacy and physical performance. This study aims to determine the effect of intradialytic aerobic exercise on improving dialysis adequacy and physical performance in twice-weekly hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* End Stage Renal Disease Patient stage 5 with Glomerular Filtration Rate <15mL/minute/1.73m2 aged 25-54 years undergoing hemodialysis two times per week for three months to five years
* Hemoglobin levels > 8mg/dl
* Mini-Mental State Examination (MMSE) score of ≥24
* Hamilton Depression Rating Scale (HDRS) score <25

Exclusion Criteria:

* Received aerobic exercise in the last 3 months
* History of hospitalization in the last 3 months
* Access for hemodialysis circulation via the femoral vein.
* IMT <18,5 (underweight) dan ≥35 (obese class II)
* Non-stable cardiovascular disease, uncontrolled glucose, acute infection disease

Ages: 25 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Kt/V | eight weeks
  Dialysis adequacy (Kt/V) and physical performance test with a Short Physical Performance Battery (SPPB) were evaluated before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Irma Ruslina Defi, Principal Investigator — Universitas Padjadjaran
Locations (1):
- Al Ihsan Hospital, Bandung, West Java, Indonesia

REFERENCES:
- [Background] Rhee SY, Song JK, Hong SC, Choi JW, Jeon HJ, Shin DH, Ji EH, Choi EH, Lee J, Kim A, Choi SW, Oh J. Intradialytic exercise improves physical function and reduces intradialytic hypotension and depression in hemodialysis patients. Korean J Intern Med. 2019 May;34(3):588-598. doi: 10.3904/kjim.2017.020. Epub 2017 Aug 25. PMID 28838226
- [Background] Yabe H, Kono K, Yamaguchi T, Ishikawa Y, Yamaguchi Y, Azekura H. Effects of intradialytic exercise for advanced-age patients undergoing hemodialysis: A randomized controlled trial. PLoS One. 2021 Oct 22;16(10):e0257918. doi: 10.1371/journal.pone.0257918. eCollection 2021. PMID 34679101